CLINICAL TRIAL: NCT02895360
Title: An Open-label Phase 1/2a Study of BAL101553 Administered as Intravenous 48-hour Infusions in Adult Patients With Advanced Solid Tumors or Recurrent Glioblastoma
Brief Title: Phase 1/2a Study of BAL101553 as 48-hour Infusions in Patients With Advanced Solid Tumors or Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDI-CS-003
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — lisavanbulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 (Experimental): Fixed 3+3 dose escalation of BAL101553 in patients with advanced solid tumors
  Interventions: Drug: BAL101553
- Phase 2a (Experimental): BAL101553 at MTD in patients with platinum-resistant/refractory ovarian cancer or recurrent glioblastoma
  Interventions: Drug: BAL101553 at MTD

INTERVENTIONS:
Drug: BAL101553 — BAL101553 48-hour infusion on day 1, 8, and 15 of each 28-day cycle; oral capsule daily for one week during Cycle 2 (study days 15-21)
  Arms: Phase 1
Drug: BAL101553 at MTD — BAL101553 48-hour infusion on day 1, 8, and 15 of each 28-day cycle; treatment with maximum tolerated dose (MTD)
  Arms: Phase 2a

SUMMARY:
Single-agent, open-label, multi-center sequential dose escalation and expansion study of BAL101553, administered as an intravenous (IV) infusion over 48 hours to adults with advanced or recurrent solid tumors or recurrent glioblastoma.

DETAILED DESCRIPTION:
This is the first study of prolonged intravenous infusion of BAL101553 (lisavanbulin). BAL101553 will be administered as an intravenous infusion over 48 hours, to adults with advanced or recurrent solid tumors or recurrent glioblastoma who have failed standard therapy, or for whom no effective standard therapy is available.

The primary goal of the study is to find the highest dose of BAL101553 that can safely be given to humans and to assess what side effects occur. The study will start by treating patients with a low dose. Once it has been shown that this low dose is well tolerated, new patients will be treated at higher dose levels ("dose escalation"). Once the highest, well tolerated dose is identified, up to 20 new patients with platinum-resistant/refractory ovarian cancer and up to 20 new patients with recurrent glioblastoma will be treated at that dose (this part is called "dose expansion") to further assess as secondary goal the tolerability and potential anticancer activity of BAL101553. A further secondary goal of this study is to assess the pharmacokinetics of BAL101553.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Phase 1: Patients with either histologically or cytologically confirmed advanced or recurrent solid tumor, who failed standard therapy or for whom no effective standard therapy is available.

   Phase 2a: Patients with platinum-resistant/refractory ovarian, fallopian tube or primary peritoneal cancer (high-grade serous, endometrioid, or carcinosarcoma histotypes) or glioblastoma in first relapse.
3. Patients with solid tumors must have measurable disease according to Response Evaluation Criteria in Solid Tumors [RECIST] v1.1.

   Patients with recurrent glioblastoma must have measurable disease defined by contrast-enhancing magnetic resonance imaging.
4. Life expectancy ≥ 12 weeks
5. Acceptable organ and marrow function at baseline (protocol defined laboratory parameters)
6. Patients with solid tumors must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 and patients with recurrent glioblastoma must have an ECOG performance status ≤ 2.
7. Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Patients with solid tumors who have received chemotherapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks prior to starting study drug or who have not recovered from side effects of prior therapies.

   Patients with recurrent glioblastoma who have: received radiotherapy within 12 weeks, unless there is a new area of enhancement consistent with recurrent tumor outside the radiation field, or there is histological confirmation of unequivocal tumor progression; received administration of prior antitumor chemotherapy within 4 weeks, or within 6 weeks for nitrosoureas; undergone surgical resection within 4 weeks or a stereotactic biopsy/core biopsy within 1 week prior to starting study drug, or have been treated previously with bevacizumab.
2. Patients who have had prior exposure to BAL101553.
3. Peripheral neuropathy ≥ CTCAE grade 2.
4. Uncontrolled intercurrent illness that would unduly increase the risk of toxicity or limit compliance with study requirements
5. Systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg at the screening visit.
6. Blood pressure (BP) combination treatment with more than two antihypertensive medications.
7. Women who are pregnant or breast-feeding. Men or women of reproductive potential who are not willing to apply effective birth control.
8. Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaindl, MD, Study Director — Basilea Pharmaceutica
Locations (6):
- Switzerland (6):
  - Oncology Institute of Southern Switzerland; Ospedale Regionale San Giovanni Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Cantonal Hospital of Grisons, Department of Oncology/ Haematology, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Cantonal Hospital of St. Gallen, Dep. Medical Oncology & Hematology, Sankt Gallen
  - UniversitaetsSpital Zürich, Zurich

REFERENCES:
- [Derived] Joerger M, Hundsberger T, Haefliger S, von Moos R, Hottinger AF, Kaindl T, Engelhardt M, Marszewska M, Lane H, Roth P, Stathis A. Safety and anti-tumor activity of lisavanbulin administered as 48-hour infusion in patients with ovarian cancer or recurrent glioblastoma: a phase 2a study. Invest New Drugs. 2023 Apr;41(2):267-275. doi: 10.1007/s10637-023-01336-9. Epub 2023 Feb 16. PMID 36792805
- [Derived] Joerger M, Stathis A, Metaxas Y, Hess D, Mantiero M, Mark M, Volden M, Kaindl T, Engelhardt M, Larger P, Lane H, Hafner P, Levy N, Stuedeli S, Sessa C, von Moos R. A Phase 1 study of BAL101553, a novel tumor checkpoint controller targeting microtubules, administered as 48-h infusion in adult patients with advanced solid tumors. Invest New Drugs. 2020 Aug;38(4):1067-1076. doi: 10.1007/s10637-019-00850-z. Epub 2019 Aug 30. PMID 31471863

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - 30 mg/m² Cohort: BAL101553 30 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 30 mg/m².
- Phase 1 - 45 mg/m² Cohort: BAL101553 45 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 45 mg/m².
- Phase 1 - 70 mg/m² Cohort: BAL101553 70 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 70 mg/m².
- Phase 1 - 90 mg/m² Cohort: BAL101553 90 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 90 mg/m².
- Phase 2a - Ovarian Cancer Cohort: BAL101553 at 70 mg/m² (MTD)
  BAL101553 as 48-hour infusion on day 1, 8, and 15 of each 28-day cycle
- Phase 2a - Recurrent Glioblastoma Cohort: BAL101553 at 70 mg/m² (MTD)
  BAL101553 48-hour infusion on day 1, 8, and 15 of each 28-day cycle
Period: Phase 1 - 30 mg/m² Cohort
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
Started | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 4 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 - 45 mg/m² Cohort
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
Started | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 3 | 0 | 0 | 0 | 0
Period: Phase 1 - 70 mg/m² Cohort
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
Started | 0 | 0 | 9 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 7 | 0 | 0 | 0
Period: Phase 1 - 90 mg/m² Cohort
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
Started | 0 | 0 | 0 | 4 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 4 | 0 | 0
Period: Phase 2a
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
Started | 0 | 0 | 0 | 0 | 11 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 11 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- 30 mg/m² Cohort: BAL101553 30 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 30 mg/m².
- 45 mg/m² Cohort: BAL101553 45 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 45 mg/m².
- 70 mg/m² Cohort: BAL101553 70 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 70 mg/m².
- 90 mg/m² Cohort: BAL101553 90 mg/m² intravenously over 48 hours on Days 1, 8 and 15 of each (at least one) 28-day treatment cycle. During cycle 2, oral BAL101553 was administered on study days 15-21. The oral dose was selected to match the weekly IV dose of 90 mg/m².
- Phase 2a - Ovarian Cancer Cohort; Phase 2a - Recurrent Glioblastoma Cohort: BAL101553 at 70 mg/m² (MTD) BAL101553 48-hour infusion on day 1, 8, and 15 of each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | 30 mg/m² Cohort | 45 mg/m² Cohort | 70 mg/m² Cohort | 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort | Total
Number analyzed (Participants) | 4 | 3 | 9 | 4 | 11 | 12 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (3.30) | 61.0 (0) | 59.6 (10.53) | 63.0 (7.26) | 64.7 (8.78) | 59.3 (7.45) | 60.7 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 6 | 3 | 11 | 3 | 27
  Male | 2 | 1 | 3 | 1 | 0 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 9 | 4 | 11 | 12 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 4 | 3 | 9 | 4 | 11 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of BAL101553
Description: First 28-day treatment cycle dose limiting toxicities (DLT) graded according to CTCAE in the MTD-determining population in Phase 1 based on the number of participants with adverse effects as measure of tolerability at various dose levels
Time Frame: 28 day cycle
Population: MTD-determining population in Phase 1: All patients who meet the following minimum criteria during the first 28-day treatment cycle (Cycle 1)
  * received at least one partial or complete dose of BAL101553 and has experienced a DLT;
  * received all three doses of BAL101553 without experiencing a DLT (including the ability to initiate treatment Cycle 2), have been observed for ≥ 28 days following the first dose, and have been evaluated for safety.
Measure: Number; unit: mg/m²
Groups:
- MTD-determining Population in Phase 1: All patients meeting the criteria of the MTD-determining population in Phase 1 during the first 28-day treatment cycle with intravenous BAL101553 at doses of 30, 45, 70 and 90 mg/m²
Arm/Group | MTD-determining Population in Phase 1
Number analyzed (Participants) | 15
mg/m² | 70

2. Secondary Outcome: Safety and Tolerability of BAL101553 Treatment Based on Number of Patients With Related Treatment-emergent Adverse Events (TEAEs) in the Phase 1 and Phase 2a Safety Population at Various Dose Levels and Indication
Description: TEAEs are defined as all events occurring after BAL101553 treatment begins, up to 28 days after last study drug administration according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Time Frame: TEAEs with onset on or after Day 1 of the study and until 28 days after the last dose
Population: All patients who receive at least one full or partial dose of BAL101553 and had at least one post-baseline safety assessment is included in the safety analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
Number analyzed (Participants) | 4 | 3 | 9 | 4 | 11 | 12
Participants
  Patients with ≥1 related AE | 2 | 2 | 8 | 3 | 9 | 4
  Patients with CTCAE Grade 3/4 or severe related AE | 0 | 0 | 2 | 2 | 3 | 1
  Patients with ≥1 related serious AE | 0 | 0 | 2 | 1 | 0 | 0

3. Secondary Outcome: AUC of BAL101553 and BAL27862
Description: Pharmacokinetic parameter "Area under the plasma concentration versus time curve" AUC0-last (of BAL101553 and BAL27862 has been assessed after a 48-hour IV infusion.
  Lisavanbulin (BAL101553) is the prodrug of avanbulin (BAL27862).
Time Frame: 0 to 168 hours post-dose at Day 1 of Cycle 1 and Cycle 2 in each cohort in Phase 1, 28-day cycles
Population: The PK analysis set includes all patients who received at least one partial or complete dose of study drug and had at least one post-baseline PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- 30 mg/m² Cycle 1 Day 1: BAL101553 30 mg/m² Cohort Cycle 1 Day 1
- 30 mg/m² Cycle 2 Day 1: BAL101553 30 mg/m² Cohort Cycle 2 Day 1
- 45 mg/m² Cycle 1 Day 1: BAL101553 45 mg/m² Cohort Cycle 1 Day 1
- 45 mg/m² Cycle 2 Day 1: BAL101553 45 mg/m² Cohort Cycle 2 Day 1
- 70 mg/m² Cycle 1 Day 1: BAL101553 70 mg/m² Cohort Cycle 1 Day 1
- 70 mg/m² Cycle 2 Day 1: BAL101553 70 mg/m² Cohort Cycle 2 Day 1
- 90 mg/m² Cycle 1 Day 1: BAL101553 90 mg/m² Cohort Cycle 1 Day 1
- 90 mg/m² Cycle 2 Day 1: BAL101553 90 mg/m² Cohort Cycle 2 Day 1
Arm/Group | 30 mg/m² Cycle 1 Day 1 | 30 mg/m² Cycle 2 Day 1 | 45 mg/m² Cycle 1 Day 1 | 45 mg/m² Cycle 2 Day 1 | 70 mg/m² Cycle 1 Day 1 | 70 mg/m² Cycle 2 Day 1 | 90 mg/m² Cycle 1 Day 1 | 90 mg/m² Cycle 2 Day 1
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 9 | 6 | 4 | 3
h*ng/mL
  BAL101553 | 1430 (43.9) | 1310 (47.6) | 2260 (43.9) | 1890 (13.3) | 3560 (45.9) | 3550 (43.1) | 4810 (74.0) | 4150 (67.5)
  BAL27862 | 1730 (37.8) | 2250 (58.2) | 3440 (45.1) | 3920 (57.7) | 7720 (44.6) | 6640 (49.3) | 10400 (37.2) | 10700 (39.3)

4. Secondary Outcome: Cmax of BAL101553 and BAL27862
Description: Pharmacokinetic parameter "Peak Plasma Concentration" Cmax of BAL101553 and BAL27862.
  Lisavanbulin (BAL101553) is the prodrug of avanbulin (BAL27862).
Time Frame: Pre-dose, and 0.5, 1, 2, 4, 8, 24, 30, 48, 52, 54, 72 h, and 168 h after the start of study-drug infusion on Day 1 of Cycle 1 and pre-dose, and 0.5, 1, 2, 4, 8, 24, 30, 48, 72 h, and 168 h after the start of study-drug infusion on Day 1 of Cycle 2.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 30 mg/m² Cycle 1 Day 1 | 30 mg/m² Cycle 2 Day 1 | 45 mg/m² Cycle 1 Day 1 | 45 mg/m² Cycle 2 Day 1 | 70 mg/m² Cycle 1 Day 1 | 70 mg/m² Cycle 2 Day 1 | 90 mg/m² Cycle 1 Day 1 | 90 mg/m² Cycle 2 Day 1
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 9 | 6 | 4 | 3
ng/mL
  BAL101553 | 43.0 (22.9) | 44.2 (15.8) | 69.3 (19.3) | 60.9 (4.3) | 119 (34.5) | 111 (34.9) | 174 (63.6) | 198 (76.8)
  BAL27862 | 45.7 (30.2) | 52.7 (45.8) | 76.8 (18.6) | 76.2 (43.1) | 144 (25.7) | 120 (41.2) | 223 (44.7) | 199 (40.4)

5. Secondary Outcome: Tmax of BAL101553 and BAL27862
Description: Pharmacokinetic parameter "Time to Peak Plasma Concentration" Tmax of BAL101553 and BAL27862
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | 30 mg/m² Cycle 1 Day 1 | 30 mg/m² Cycle 2 Day 1 | 45 mg/m² Cycle 1 Day 1 | 45 mg/m² Cycle 2 Day 1 | 70 mg/m² Cycle 1 Day 1 | 70 mg/m² Cycle 2 Day 1 | 90 mg/m² Cycle 1 Day 1 | 90 mg/m² Cycle 2 Day 1
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 9 | 6 | 4 | 3
hours
  BAL101553 | 39.0 [24.0 to 48.0] | 30.0 [24.0 to 48.0] | 29.0 [4.03 to 30.0] | 27.1 [24.2 to 30.0] | 4.00 [1.00 to 24.1] | 1.56 [1.00 to 4.05] | 2.53 [1.03 to 46.5] | 1.17 [1.00 to 3.95]
  BAL27862 | 48.0 [30.1 to 48.0] | 48.0 [24.0 to 52.9] | 48.0 [29.0 to 48.1] | 47.5 [47.2 to 47.9] | 47.6 [29.1 to 52.1] | 46.6 [7.5 to 54.7] | 46.2 [23.8 to 47.5] | 47.4 [46.7 to 47.4]

6. Secondary Outcome: Bioavailability of Daily Oral BAL101553 Measured by BAL27862 in Phase 1
Description: Ratio of AUCs of avanbulin after oral and IV administration (relative bioavailability) of BAL101553 (lisavanbulin) which is the prodrug of avanbulin (BAL27862)
Time Frame: Relative oral bioavailability, calculated as dose-normalized AUC0-τ following oral administration on Cycle 2 Day 21 divided by dose normalized AUC0-∞ following IV administration on Cycle 1 Day 1 for each cohort.
Population: Patients with both Cycle 1 Day 1 AUC0-∞ and Cycle 2 Day 1 AUC0-τ evaluations
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- 30 mg/m²; 45 mg/m²; 70 mg/m²; 90 mg/m²: Patients with both Cycle 1 Day 1 AUC0-∞ and Cycle 2 Day 1 AUC0-τ evaluations
Arm/Group | 30 mg/m² | 45 mg/m² | 70 mg/m² | 90 mg/m²
Number analyzed (Participants) | 1 | 1 | 3 | 1
Ratio | 1.11 (0) | 1.32 (0) | 0.796 (18.9) | 0.893 (0)

7. Secondary Outcome: Anti-tumor Activity of BAL101553 by Best Response Rate Per RECIST / RANO Criteria
Description: The objective response rate (ORR) was calculated using the efficacy evaluable populations (EEPs in Phase 2a) and the full analysis population (FAP in Phase 1 and Phase 2a) based on RECIST v1.1 guidelines (defines criteria for the radiological assessment in tumor response) for patients with solid tumors (excluding GBM (glioblastoma)) and RANO criteria (assessment Incorporating MRI and clinical factors) for patients with GBM.
  ORR = Rate of complete and partial responses
Time Frame: 28 day cycles
Population: FAP:
  Patients who receive at least one partial or complete dose of BAL101553.
  EEP:
  Patients with progressive disease who completed at least Cycle 1 dosing and at least one on-study tumor assessment (clinical or radiological by RECIST v1.1 or RANO criteria) Patients with stable disease, partial or complete response, based on a radiological assessment by RECIST v1.1 or RANO criteria at the end of Cycle 2, with at least 4 doses of study drug in the first two cycles.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1- in the FAP: All dose cohorts (30 mg/m², 45 mg/m², 70 mg/m² and 90 mg/m²) of BAL101553 in patients with advanced solid tumors
  BAL101553 48-hour infusion on day 1, 8, and 15 of each 28-day cycle; oral capsule daily for one week during Cycle 2
- Phase 2a - Patients With Ovarian Cancer in the FAP; Phase 2a - Patients With Ovarian Cancer in the EEP; Phase 2a - Patients With Recurrent Glioblastoma in the FAP; Phase 2a - Patients With Recurrent Glioblastoma in the EEP: BAL101553 at 70 mg/m² (MTD)
  BAL101553 48-hour infusion on day 1, 8, and 15 of each 28-day cycle
Arm/Group | Phase 1- in the FAP | Phase 2a - Patients With Ovarian Cancer in the FAP | Phase 2a - Patients With Ovarian Cancer in the EEP | Phase 2a - Patients With Recurrent Glioblastoma in the FAP | Phase 2a - Patients With Recurrent Glioblastoma in the EEP
Number analyzed (Participants) | 20 | 11 | 8 | 12 | 8
Participants
  Complete response | 1 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 1 | 1
  Stable disease | 3 | 4 | 3 | 2 | 1
  Progressive disease | 15 | 7 | 5 | 9 | 6
  Missing | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug through 28 days after the administration of the last dose
Description: TEAEs with onset on or after Day 1 of the study and until 28 days after the last dose.
Arm/Group | Phase 1 - 30 mg/m² Cohort | Phase 1 - 45 mg/m² Cohort | Phase 1 - 70 mg/m² Cohort | Phase 1 - 90 mg/m² Cohort | Phase 2a - Ovarian Cancer Cohort | Phase 2a - Recurrent Glioblastoma Cohort
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 3/9 | 0/4 | 3/11 | 2/12
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 7/9 | 1/4 | 4/11 | 5/12
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 9/9 | 4/4 | 11/11 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - 30 mg/m² Cohort (N=4) | Phase 1 - 45 mg/m² Cohort (N=3) | Phase 1 - 70 mg/m² Cohort (N=9) | Phase 1 - 90 mg/m² Cohort (N=4) | Phase 2a - Ovarian Cancer Cohort (N=11) | Phase 2a - Recurrent Glioblastoma Cohort (N=12)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - 30 mg/m² Cohort (N=4) | Phase 1 - 45 mg/m² Cohort (N=3) | Phase 1 - 70 mg/m² Cohort (N=9) | Phase 1 - 90 mg/m² Cohort (N=4) | Phase 2a - Ovarian Cancer Cohort (N=11) | Phase 2a - Recurrent Glioblastoma Cohort (N=12)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Hemianaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurologic neglect syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (7) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (4) | 6 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 6 (7) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 3 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (4) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (5) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (7) | 3 (3) | 6 (6) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 3 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 8 (9) | 3 (5) | 6 (14) | 4 (4)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 1 (1) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 4 (7) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02895360/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT02895360/SAP_001.pdf